CLINICAL TRIAL: NCT06683742
Title: A 2-year Phase 3, Multicenter, Prospective, Randomized, Double-Masked, Parallel-Group Study of EYP-1901, a Tyrosine Kinase Inhibitor (TKI), Compared to Aflibercept in Subjects With Wet AMD
Brief Title: A 2-year Study of EYP-1901 in Subjects With Wet Age Related Macular Degeneration (wAMD) (LUCIA) Primary Efficacy Will be Determined at Week 56
Acronym: wAMD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EYP-1901-302
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Wet Age Related Macular Degeneration; wAMD
Keywords: Wet Age-related Macular Degeneration; Tyrosine Kinase Inhibitor; EYP-1901; EyePoint
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EYP-1901 2686 µg (Experimental): EYP-1901
  Interventions: Drug: EYP-1901
- Aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept (2.0 mg)

INTERVENTIONS:
Drug: EYP-1901 — Intravitreal Injection
  Arms: EYP-1901 2686 µg
Drug: Aflibercept (2.0 mg) — Intravitreal Injection
  Arms: Aflibercept

SUMMARY:
This is a phase 3 randomized, double -masked study comparing the efficacy of EYP-1901 against Aflibercept.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated or treatment naïve patients with a documented diagnosis of wAMD in the study eye, with onset of disease that began at any time prior to the Screening Visit.
* Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) letter score between 78 to 35 letters (approximately 20/32 to 20/200 Snellen equivalent) in the study eye at the Screening Visit and on Baseline (Day 1).
* For previously-treated subjects, must have been treated with at least 2 anti-VEGF IVT injections (i.e., aflibercept 2 mg, aflibercept 8 mg, bevacizumab, ranibizumab, or faricimab) in the previous 6 months for wAMD per standard of care in the study eye prior to the Screening Visit.

Exclusion Criteria:

* Subfoveal fibrosis, atrophy, or scarring in the center subfield.
* BCVA using ETDRS charts <20 letters (20/400 Snellen equivalent) in the fellow eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Average change in best corrected visual acuity (BCVA) | Weeks 52 and 56

SECONDARY OUTCOMES:
Rate of injection burden | Week 56
Average change in best corrected visual acuity (BCVA) | Week 96

CONTACTS AND LOCATIONS:
Locations (150):
- United States (106):
  - Associated Retina Consultans, Gilbert, Arizona
  - Associated Retina Consultants - Phoenix, Phoenix, Arizona
  - Phoenix Retina Clinical Trials, LLC, Phoenix, Arizona
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - Win Retina, Arcadia, California
  - Doctor Retina, PC, Beverly Hills, California
  - The Retina Partners, Encino, California
  - RCOC Clinical Research Institute Inc., Fullerton, California
  - Global Research Management, Inc., Glendale, California
  - Atlantis Eyecare, Huntington Beach, California
  - South Coast Retina Center, Long Beach, California
  - Retinal Consultants Medical Group, Modesto, California
  - Northern California Retina Vitreous Associates Medical Group INC., Mountain View, California
  - Kaiser Permanente, Oakland, California
  - California Retina Consultants Oxnard Office, Oxnard, California
  - Retina Consultants San Diego, Poway, California
  - California Eye Specialists Medical Group, Inc., Redlands, California
  - Retina Consultants of Southern California, Redlands, California
  - SCPMG/Kaiser Permanente Riverside Medical Center, Riverside, California
  - VRMG Inc, Sacramento, California
  - Retinal Consultants Medical Group, Sacramento, California
  - West Coast Retina Medical Group, San Francisco, California
  - Macula Retina Vitreous Research Institute, Torrance, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - RSC Research, PLLC, Denver, Colorado
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Colorado Retina Associates, Lakewood, Colorado
  - Connecticut Eye Consultants, P.C., Danbury, Connecticut
  - SightSera Clinical Research LLC, Greenwich, Connecticut
  - Retina Group of New England, PC, Waterford, Connecticut
  - Blue Ocean Clinical Research, Clearwater, Florida
  - Advanced Research, LLC, Deerfield Beach, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - The Eye Institute of West Florida, Largo, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - MedEye Associates, South Miami, Florida
  - Retina Vitreous Associates of Florida - Saint Petersburg, St. Petersburg, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Retina Specialists of Tampa, Tampa, Florida
  - Georgia Retina, Marietta, Georgia
  - Gailey Eye Clinic, Bloomington, Illinois
  - Retina Associates, Elmhurst, Illinois
  - Illinois Retina Associates, S.C., Oak Park, Illinois
  - Red River Research Partners, Plainfield, Illinois
  - AVRUC, Carmel, Indiana
  - Retina Associates of Kentucky, Lexington, Kentucky
  - The Eye Care Institute, Louisville, Kentucky
  - Retina Associates New Orleans, Metairie, Louisiana
  - Haik Humble Eye Center, West Monroe, Louisiana
  - The Retina Care Center, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - Discover Vision Center, Independence, Missouri
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Mid Atlantic Retina, Cherry Hill, New Jersey
  - NJ Retina, Edison, New Jersey
  - NJ Retina, Toms River, New Jersey
  - Retina Vitreous Surgeons of CNY, PC, Liverpool, New York
  - NYC Retina, New York, New York
  - Retina Associates of Western NY, PC, Rochester, New York
  - VRCNY/Long Island Vitreoretinal Consultants, Westbury, New York
  - NC Retina Associates - Cary Research, Cary, North Carolina
  - Graystone Eye - Hickory Office, Hickory, North Carolina
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Retina Vitreous Center, PLLC, Edmond, Oklahoma
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Casey Eye Institute at OHSU, Portland, Oregon
  - Cascade Medical Research lnstitute, LLC, Springfield, Oregon
  - Wills Eye Physician Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Erie Retina Research, Erie, Pennsylvania
  - Retina Vitreous Consultants (RVC) - Monroeville, Monroeville, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Tennessee Retina, Nashville, Tennessee
  - Panhandle Eye Group, LLP. - Southwest Retina Specialists, Amarillo, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - TX RCTX Retina Consultants of Texas, Beaumont, Texas
  - Star Vision Research, Burleson, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina of North Texas, Dallas, Texas
  - Berkeley Eye Center, Houston, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Valley Retina Institute P.A., McAllen, Texas
  - Red River Research Partners, LLC, Plano, Texas
  - Texas Retina Associates, Plano, Texas
  - TX RCTX Retina Consultants of Texas, San Antonio, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Retina Associates of South Texas, San Antonio, Texas
  - Tyler Retina Consultants, Tyler, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Salt Lake Retina, West Jordan, Utah
  - The Retina Group of Washington, Fairfax, Virginia
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia
  - Virginia Retina Center, Warrenton, Virginia
  - Pacific Northwest Retina, Bellevue, Washington
- Australia (3):
  - Eye Clinic Albury Wodonga, Albury
  - Marsden Eye Specialists, Parramatta
  - Sydney Retina Clinic and Day Surgery, Sydney
- Brazil (6):
  - Retina Prime at Jardim Europa Medical Center, Aracaju
  - Centro Brasileiro de Pesquisa Clinica - Blumenau, Blumenau
  - Clínica Oftalmológica São Lucas - Retina Clinic, São Paulo
  - Hospital de Olhos Oeste Paulista, São Paulo
  - UNIFESP - Hospital Sao Paulo, São Paulo
  - Hospital Oftalmológico de Sorocaba (Centro de Estudos), Sorocaba
- Czechia (3):
  - VISUS, spol s.r.o., Náchod
  - Axon Clinical, s.r.o., Prague
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- St Elisabeth Krankenhaus, Cologne, Germany
- Hungary (5):
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Budapest Retina Associates, Budapest
  - Debreceni Egyetem KK Szemklinika, Debrecen
  - Ganglion Medical Center, Pécs
  - Pecsi Tudomanyegyetem AOK, Pécs
- India (8):
  - Rising Retina Clinic, Ahmedabad
  - Narayana Netralaya, Bengaluru
  - Netralayam VIP, Kolkata
  - Aravind Eye Hospital and Postgraduate Institute of Ophthalmology, Madurai
  - Shanti Saroj Netralay, Miraj
  - K. B. Haji Bachooali Charitable Ophthalmic & E.N.T. Hospital, Mumbai
  - Shroff Eye Hospital, Mumbai
  - Netrodaya - The Eye City, Varanasi
- Israel (8):
  - Shamir Medical Center Ophthalmology Out Patient Clinic, Be’er Ya‘aqov
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Meir Medical Center Ophthalmology Department, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - The Tel-Aviv Sourasky Medical Centre, Tel Aviv
- Poland (7):
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Szpital sw. Rozy- obsolete; New Name: Szpital Św. Róży sp. z o.o., Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Centrum Diagnostyki i Mikrochirurgii Oka -LENS Sp. z o. o, Olsztyn
  - Centrum Medyczne UNO-MED, Tarnów
  - Piasta 47 Centrum Medyczne, Warsaw
  - Warszawski Szpital Okulistyczny, Warsaw
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta Banska Bystrica, Banská Bystrica
  - CMO Bratislava, Bratislava
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided